CLINICAL TRIAL: NCT05555667
Title: Long-term Sedation With Remimazolam Besylate Versus Propofol in Critically Ill Patients During Invasive Mechanical Ventilation: a Randomized Non-inferior Trial
Brief Title: Long-term Sedation With Remimazolam Besylate in Critically Ill Patients
Acronym: LOSREB
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xiaobo Yang, MD, Clinical Professor, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WHUICU202209
Record Dates: First submitted 2022-09-22; First posted 2022-09-27 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2022-09

CONDITIONS: Light Sedation; Mechanical Ventilation
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remimazolam besylate (Experimental): Remimazolam besylate at an initial infusion rate of 0.15 mg/kg/h and adjusted (maximum of 0.3 mg/kg/h) to maintain a RASS score between - 3 and 0
  Interventions: Drug: Remimazolam besylate
- Propofol (Active Comparator): Propofol intravenously at an initial infusion rate of 2.0 mg/kg/h and adjusted (maximum of 4.0 mg/kg/h) to maintain a RASS score between - 3 and 0
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Remimazolam besylate — Sedation drug
  Arms: Remimazolam besylate
Drug: Propofol — Propofol. Sedation drug
  Arms: Propofol

SUMMARY:
A randomized non-inferior trial comparing remimazolam besylate with propofol for long-term sedation during invasive mechanical ventilation in critically ill patients

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤ 80 years;
* Intubated and mechanically ventilated ≤96 hours before enrollment；
* Expected to require continuous invasive ventilation and sedation ≥24 hours;
* Requirement for light to moderate sedation (a RASS score of -3 to 0)

Exclusion Criteria:

* Body mass index (BMI) <18 or >30 kg/m2;
* Allergy or unsuitabilty to any composition of study drugs or remifentanil;
* Living expectancy less than 48 hours；
* Possible surgey in the operating room in 24 hours；
* Myasthenia gravis;
* Serious hepatic dysfunction (CTP 10-15);
* Chronic kidney disease with glomerular filtration rate (GFR) < 29 ml/min/1.73m2;
* Systolic blood pressure less than 90 mm Hg after appropriate intravenous volume replacement and continuous infusions of 2 vasopressors;
* Acute severe neurological disorder and any other condition interfering with RASS assessment;
* Pregnancy or lactation;
* Unstable angina or acute myocardial infarction;
* Left ventricular ejection fraction less than 30%;
* Heart rate less than 50 beats/min;
* Grade 2 , second degree or third degree atrioventricular block in the absence of a pacemaker;
* Abuse of controlled substances or alcohol;
* Other conditions deemed unsuitable to be included;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 728 (Estimated)
Dates: Start 2023-05-16 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
The percentage of time in the target sedation range without rescue sedation | 7 days after enrollment, or when patients decease, require deep sedation, are scheduled for surgery, are discontinued from the study drug for at least 12 hours, are discharged from ICU, or are withdrawn from the trial, whichever comes first
  The percentage of time in the target sedation range without rescue sedation

SECONDARY OUTCOMES:
Invasive ventilator free time | From start of study to 7 days
  Hours of time free from invasive ventilator
Successful extubation rate | From start of study to 7 days
  Extubation of endotracheal tube for the first time in 7 days without reintubation or switching to tracheostomy within the following 48 hours
Length of ICU stay | From start of study to 28 days
  Length of ICU stay
Mortality | From start of study to 28 days
  Mortality
Length of hospitalization | From start of study to 28 days
  Length of hospitalization
weaning time | From start of study to 7 days
  weaning time in minutes between continuous discontinuation of the study drug and extubation in patients with successful extubation
Rate of hypotension | 7 days after enrollment, or when patients decease, require deep sedation, are scheduled for surgery, are discontinued from the study drug for at least 12 hours, are discharged from ICU, or are withdrawn from the trial, whichever comes first
  Systolic blood pressure less than 80 mmHg or diastolic blood pressure less than 50 mmHg for 5 minutes or treated with vasopressors
Rate of hypertension | 7 days after enrollment, or when patients decease, require deep sedation, are scheduled for surgery, are discontinued from the study drug for at least 12 hours, are discharged from ICU, or are withdrawn from the trial, whichever comes first
  systolic blood pressure greater than 160 mm Hg or diastolic blood pressure greater than 100 mmHg for 5 minutes or treated with vasodilators
Rate of bradycardia | 7 days after enrollment, or when patients decease, require deep sedation, are scheduled for surgery, are discontinued from the study drug for at least 12 hours, are discharged from ICU, or are withdrawn from the trial, whichever comes first
  heart rate less than 50 bpm for 5 minutes or treated with medication to increase heart rate
Rate of tachycardia | 7 days after enrollment, or when patients decease, require deep sedation, are scheduled for surgery, are discontinued from the study drug for at least 12 hours, are discharged from ICU, or are withdrawn from the trial, whichever comes first
  heart rate greater than 120 bpm for 5 minutes or treated with medication to decrease heart rate
Rate of unplanned extubation of endotracheal tube | 7 days after enrollment, or when patients decease, require deep sedation, are scheduled for surgery, are discontinued from the study drug for at least 12 hours, are discharged from ICU, or are withdrawn from the trial, whichever comes first
  unplanned extubation of endotracheal tube
Rate of shock | 7 days after enrollment, or when patients decease, require deep sedation, are scheduled for surgery, are discontinued from the study drug for at least 12 hours, are discharged from ICU, or are withdrawn from the trial, whichever comes first
  New-onset shock
Rate of hospital-acquired pneumonia | 7 days after enrollment, or when patients decease, require deep sedation, are scheduled for surgery, are discontinued from the study drug for at least 12 hours, are discharged from ICU, or are withdrawn from the trial, whichever comes first
  hospital-acquired pneumonia
Rate of myocardial infarction | 7 days after enrollment, or when patients decease, require deep sedation, are scheduled for surgery, are discontinued from the study drug for at least 12 hours, are discharged from ICU, or are withdrawn from the trial, whichever comes first
  myocardial infarction
Rate of cerebral ischemic stroke | 7 days after enrollment, or when patients decease, require deep sedation, are scheduled for surgery, are discontinued from the study drug for at least 12 hours, are discharged from ICU, or are withdrawn from the trial, whichever comes first
  cerebral ischemic stroke
Rate of cerebral hemorrhagic stroke | 7 days after enrollment, or when patients decease, require deep sedation, are scheduled for surgery, are discontinued from the study drug for at least 12 hours, are discharged from ICU, or are withdrawn from the trial, whichever comes first
  Rate of cerebral hemorrhagic stroke
Rate of pulmonary embolism | 7 days after enrollment, or when patients decease, require deep sedation, are scheduled for surgery, are discontinued from the study drug for at least 12 hours, are discharged from ICU, or are withdrawn from the trial, whichever comes first
  pulmonary embolism
Rate of upper digestive tract ulcer confirmed endoscopically | 7 days after enrollment, or when patients decease, require deep sedation, are scheduled for surgery, are discontinued from the study drug for at least 12 hours, are discharged from ICU, or are withdrawn from the trial, whichever comes first
  upper digestive tract ulcer confirmed endoscopically
Rate of more than 500 milliliters of bloody stool | 7 days after enrollment, or when patients decease, require deep sedation, are scheduled for surgery, are discontinued from the study drug for at least 12 hours, are discharged from ICU, or are withdrawn from the trial, whichever comes first
  more than 500 milliliters of bloody stool
Rate of delirium | 7 days after enrollment, or when patients decease, require deep sedation, are scheduled for surgery, are discontinued from the study drug for at least 12 hours, are discharged from ICU, or are withdrawn from the trial, whichever comes first
  delirium
delta SOFA | 7 days after enrollment, or when patients decease, require deep sedation, are scheduled for surgery, are discontinued from the study drug for at least 12 hours, are discharged from ICU, or are withdrawn from the trial, whichever comes first
  defined as the difference between SOFA when each patient stops receiving the study drug and SOFA at inclusion
Rate of withdraw from the trial because of intolerance, severe adverse events or other safety concerns | 7 days after enrollment, or when patients decease, require deep sedation, are scheduled for surgery, are discontinued from the study drug for at least 12 hours, are discharged from ICU, or are withdrawn from the trial, whichever comes first
  rate of withdraw from the trial because of intolerance, severe adverse events or other safety concerns

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Critical Care Medicine, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yang X, Tang Y, Du R, Yu Y, Xu J, Zhang J, Liu H, Zou X, Ren L, Yuan S, Shang Y. Long-term sedation with remimazolam besylate versus propofol in critically ill patients during invasive mechanical ventilation: a study protocol for a multicenter randomized non-inferior trial. Front Pharmacol. 2023 Jul 28;14:1139872. doi: 10.3389/fphar.2023.1139872. eCollection 2023. PMID 37576823